CLINICAL TRIAL: NCT04075708
Title: First Trimester Screening for Late-onset Preeclampsia: Evaluation of Novel Predictive Biomarker MMP-7 in Combination With MAP and Uterine Artery Pulsatility Index in a Danish Population
Brief Title: Predicting Late-onset Preeclampsia at 10-14 Weeks of Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-031 PIKBF PRESIDE
Record Dates: First submitted 2019-08-23; First posted 2019-09-03 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-11

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 0.5 mL serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-group: The case group will consist of women diagnosed with PE after 34 weeks of gestation.
- Control-group: The control group will include 165 participants who were not diagnosed with PE in their pregnancies.

SUMMARY:
The aim of this study is to make it easier to predict late-onset preeclampsia at 11-14 weeks of pregnancy. This will be done by measuring certain proteins in the mother's blood together with obtaining the mother's medical history, ultrasound of the mother's blood supply to the uterus, and her blood pressure.

All expectant mothers who meet the inclusion criteria will be invited to participate in the study, and those that agree will have the above mentioned factors measured at their first trimester scan appointment. The data will be registered in an online database, and the blood samples will be saved in a biobank at the hospital.

When the women have then given birth around six months later, the data will be analyzed, and whether or not the individual woman ended up developing preeclampsia will be found out from her medical records. It will then be possible to see if blood samples, medical history, blood supply to the uterus, and/or blood pressure are connected to development of preeclampsia.

DETAILED DESCRIPTION:
The aim of this study is to improve the current first-trimester screening regimes for early detection of late-onset preeclampsia (PE) using maternal serum biomarkers in combination with maternal history, uterine artery flow, and mean arterial blood pressure.

Hypothesis: Matrix metalloproteinase 7 (MMP-7) in combination with maternal history, uterine artery flow and mean arterial blood pressure can improve the detection rate of late onset PE.

The Fetal Medicine Foundation (FMF) algorithm is developed with the objective of identifying women at high risk of PE in the first trimester of pregnancy, allowing for effective prophylactic use of low-dose acetylsalicylic acid (ASA) started before 16 weeks of pregnancy. The algorithm utilizes Bayes' theorem by combining maternal characteristics and medical history with uterine artery pulsatility index (PI), mean arterial pressure (MAP), maternal serum pregnancy-associated plasma protein-A (PAPP-A), and placental growth factor (PlGF) and has been validated in several populations. It has been shown to identify up to 90% of early-onset PE (EO-PE) cases, however, the detection rate of late-onset PE (LO-PE) remains low and the biomarkers PAPP-A and PlGF do not appear to significantly improve performance of screening for these cases compared to screening by maternal characteristics and medical history alone.

An abundance of biomarkers have been suggested and researched for the prediction of LO-PE and of these, matrix metalloproteinase 7 (MMP-7) has shown to be a potentially useful predictor with a sensitivity of 69% at a false positive rate (FPR) 20% at 8-16 weeks of pregnancy. Additionally, MAP appears to be a relatively good predictor for LO-PE at the same gestational age (GA). Ultimately, the search for more accurate biomarkers and prediction models for PE and especially for LO-PE remains relevant and necessary, both with regards to improving antenatal care and taking the necessary precautions for PE mothers, researching potential treatments, and gaining a better understanding of PE pathophysiology altogether.

This study will be a nested case-control study carried out as a sub-study of the larger multicenter study "Preeclampsia Screening in Denmark" (PRESIDE) comprising six major hospitals in Denmark, including Odense University Hospital (OUH). Throughout the time period September 2019 to March 2020, 1400 participants are expected to enroll in PRESIDE through OUH with the goal of validating the FMF screening algorithm in a Danish population. These women will be giving birth from March to June 2020. In our sub-study, the case group will consist of women diagnosed with PE after 34 weeks of gestation. With an expected late-onset PE incidence of 2,5%, the sample size of the case group will be n=35. The control group will include 165 participants who were not diagnosed with PE in their pregnancies.

All information regarding maternal characteristics and medical history are collected as part of standard procedure during first trimester screening for chromosomal abnormalities and is stored in theOUH fetal medicine database Astraia. Uterine artery flow values will be entered in Astraia along with these data. Mean arterial pressure (MAP) measurements will be automatically transferred to a REDCap database where all study data, including consent forms and outcome data, will be stored. For all participants, information regarding pregnancy and neonatal outcome will be collected from registers and individual patient files. The collected blood samples will be stored and analyzed after the child is born and hence, the PE risk will only be calculated after delivery. Venous blood will be sampled, and aliquots will be stored as part of a research biobank and a biobank for future research at the Department of Clinical Biochemistry and Pharmacology (KBF), OUH. The samples for measurement of MMP-7 will be taken from the biobank for future research and will be performed in the Biomarker Laboratory at the KBF research unit by an automated immunoassay analyzer system (Tritius) using a Human Total MMP-7 Quantikine ELISA Kit.

The cohort consists of pregnant women assigned to the Department of Obstetrics at Odense University Hospital for their first trimester nuchal translucency between September 2019 and March 2020; who are included/excluded according to the criteria; and who agree to enroll in the study. The potential participants will receive information about the study by e-boks (online communication platform) when they book their appointment for the first trimester scan and will be approached by project staff upon arrival to the department on the day of the scan. Those who agree to receive more information will be orally informed by project staff about the project and its implications. Each participant will provide written consent followed by blood sampling, MAP measurements, and ultrasound procedures.

ELIGIBILITY:
Inclusion Criteria:

* A planned first trimester nuchal translucency scan
* Informed consent
* Gestational age 11-14 weeks at the first trimester scan

Exclusion Criteria:

* Age < 18 years
* ≥ 2 fetuses
* Participants must read and understand Danish or English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort consists of pregnant women assigned to the Department of Obstetrics at Odense University Hospital for their first trimester nuchal translucency between September 2019 and March 2020; who are included/excluded according to the criteria below; and who agree to enroll in the study.
Sampling Method: Probability Sample
Enrollment: 1427 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Late-onset preeclampsia | After delivery of the child, i.e. an average of 6 months from enrollment
  Diagnosis of pre-eclampsia >34 weeks of pregnancy

SECONDARY OUTCOMES:
Fetal growth restriction | After delivery of the child, i.e. an average of 6 months from enrollment
  Neonates born with a birthweight < -21% or with signs of adaption to undernutrition
Gestational hypertension | After delivery of the child, i.e. an average of 6 months from enrollment
  Women who experienced new-onset hypertension in their pregnancies
Apgar score | After delivery of the child, i.e. an average of 6 months from enrollment
  Apgar scores of neonates born to the cohort
Method of delivery | After delivery of the child, i.e. an average of 6 months from enrollment
  Method of delivery (i.e. vaginal, elective Cesarean, emergency Cesarean) in the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Lene Sperling, M.D., PhD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

DOCUMENTS (1):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT04075708/Prot_002.pdf